CLINICAL TRIAL: NCT06154967
Title: To Explore the Effect of Immune-induced Stereotactic Body Radiotherapy (SBRT) on Reversing Immunoresistance in Stage IIIc/IV Non-small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Xiong Yanli, MD, Associate Medical Director, Oncology, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DPCC-20231122
Record Dates: First submitted 2023-11-23; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Non-Small Cell Lung Cancer Without Mutation in Epidermal Growth Factor Receptor (Disorder)
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ICIs regimen: tislelizumab 200mg every 3 weeks, the first dose was given 7 days after the last SBRT (Experimental)
  Interventions: Radiation: tereotactic body radiotherapy

INTERVENTIONS:
Radiation: tereotactic body radiotherapy — In second-line and later treatment, the treatment regimen of SBRT combined with tislelizumab is used
  Other Names: tislelizumab

SUMMARY:
The goal of this clinical trial is to learn about in describe participant population. The main questions it aims to answer are:

the outcomes of the efficacy (ORR) and safety (adverse events, including irAEs, AE, SAEs, and laboratory indicators) of continued immunotherapy in patients with immune-resistant IIIc/IV metastatic NSCLC treated with immune-induced radiotherapy (SBRT).

Participants will be asked to accept the treatment of ICIs regimen and SBRT plan as follows:

ICIs regimen: tislelizumab 200mg every 3 weeks, the first dose was given 7 days after the last SBRT treatment, then the first day of each cycle, 21 days as a cycle until disease progression.

SBRT plan: The radiation dose and fractionation of SBRT should be evaluated according to the size and location of the tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with IIIc/IV NSCLC confirmed by histology and imaging
2. Previous treatment with anti-PD1 or anti-PDL1, and resistantance to ICIs
3. Without standard treatment regimen
4. At least one measurable target (primary tumour or metastasis) according to RECIST v1.1
5. Age ≥ 18 and ≤ 75
6. ECOG PS ≤ 2
7. Life expectancy ≥ 3 months

Exclusion Criteria:

1. Autoimmune disease that might be aggravated during treatment with an immuno-stimulating agent (patients with type I diabetes, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible)
2. Immunosuppressive long-term treatment (patients necessitating a corticotherapy are eligible if they are administered in doses < or = to the equivalent of 10 mg of prednisone daily, administration of steroids by a route resulting in minimal systemic exposure (local, intra-anal, intraocular or inhalation) are eligible).
3. Transplant patients (including stem cell transplants), HIV positive or other immune deficiency syndromes
4. Active infection by HBV or HCV Known severe hypersensitivity to monoclonal antibodies or history of anaphylactic shock, or uncontrolled asthma
5. Patient with interstitial pneumonitis or pulmonary fibrosis or any other known severe respiratory insufficiency
6. Patient already included in another clinical trial during treatment with an experimental

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The Overall Response Rate out of the radiation field | Individual patients should be evaluated within 3 days after the patient follow-up examination
  To evaluate the efficacy of this protocol，Measurements were based on recist1.1